CLINICAL TRIAL: NCT07191483
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, Pharmacokinetics (PK), and Pharmacodynamics (PD) of KYN-5356 as Adjunctive Treatment in Adults With Cognitive Impairment Associated With Schizophrenia
Brief Title: A Study to Evaluate KYN-5356 in Adults With Cognitive Impairment Associated With Schizophrenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kynexis B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KYN5356-CL-002
Record Dates: First submitted 2025-09-10; First posted 2025-09-24 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Impairment Associated With Schizophrenia (CIAS)
Keywords: Schizophrenia; Cognitive Dysfunction
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- KYN-5356 low dose (Experimental): KYN-5356 low dose, oral tablet for 28 days
  Interventions: Drug: KYN-5356 low dose
- KYN-5356 medium dose (Experimental): KYN-5356 medium dose, oral tablet for 28 days
  Interventions: Drug: KYN-5356 Medium Dose
- KYN-5356 high dose (Experimental): KYN-5356 high dose, oral tablet for 28 days
  Interventions: Drug: KYN-5356 High Dose
- Placebo (Placebo Comparator): Placebo, oral tablet for 28 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: KYN-5356 low dose — oral tablet
  Arms: KYN-5356 low dose
Other: Placebo — Oral tablet
  Arms: Placebo
Drug: KYN-5356 Medium Dose — oral tablet
  Arms: KYN-5356 medium dose
Drug: KYN-5356 High Dose — oral tablet
  Arms: KYN-5356 high dose

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled study to evaluate the efficacy, safety, Pharmacokinetic (PK) and Pharmacodynamic (PD) effects of 3 different dose regiments of KYN-5356 and placebo for 28 days.

Participants will be randomized to one of 4 treatment groups: placebo, KYN-5356 low dose, KYN-5356 medium dose, KYN-5356 high dose.

Participants will be admitted to the clinic on Day -3 and will remain in residence at the clinic for 32 days, from baseline through the treatment period.

Participants will be administered investigational medicinal product on Days 1 through 28. Efficacy, safety, PK and exploratory PD assessments will be performed throughout the dosing period. Participants will be discharged on Day 29 after safety assessments are completed and return for a follow-up visit on Day 42.

A subset of participants from selected sites will undergo electrophysiological assessments to evaluate the effect of KYN-5356 on neurophysiological measures of brain function.

ELIGIBILITY:
Inclusion Criteria:

* Has an established primary psychiatric diagnosis of schizophrenia
* Clinically stable and in the residual (nonacute) phase of their illness for at least 8 weeks before screening in the judgement of the investigator
* Diagnosis of schizophrenia for at least 1 year before screening
* Must be in ongoing maintenance antipsychotic monotherapy on a stable medication treatment regimen for ≥ 2 months before screening, including concomitant psychotropic medications.
* Male or female, aged ≥18 and ≤55 years
* Has a body mass index (BMI) between 18 and 40 kg/m2 Inclusive
* Must exhibit capability to comply with all protocol procedures in the judgement of the investigator
* Signed and dated written informed consent before screening in accordance with Good Clinical Practice.

Exclusion Criteria:

* Currently being treated with more than 1 antipsychotic at the time of screening,
* A score of 2 or higher on any of the individual items of the Modified Simpson-Angus Scale (mSAS) at screening
* Moderate to severe substance use disorder (other than nicotine or caffeine, but including alcohol)
* Evidence of unstable medical condition

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of KYN-5356 treatment on cognitive function in adults with cognitive impairment associated with schizophrenia (CIAS) | 28 days
  Change from Baseline at Day 28 in the digital version of the Brief Assessment of Cognition for Schizophrenia (BAC App) composite T-score

SECONDARY OUTCOMES:
Cmax | 28 days
  Maximum concentration (Cmax) of KYN-5356 and relevant KYN-5356 metabolites on Day 1 and Day 28
AUCtau | 28 Days
  Area under the concentration-time curve from time 0 to tau (end of dosing interval) (AUCtau) of KYN-5356 and relevant KYN-5356 metabolites on Day1 and Day 28
Tmax | 28 Days
  Time to Cmax (Tmax) of KYN-5356 and relevant KYN-5356 metabolites on Day1 and Day 28
Ctrough | 28 Days
  Trough concentration (Ctrough) of KYN-5356 and relevant KYN-5356 metabolites on Days 1, 7, 14, 21, and 28
Terminal half-life (t1/2) | 28 Days
  Terminal half-life (t1/2) after the last dose on Day 28 for KYN-5356 and relevant KYN-5356 metabolites

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Woodland International Research Group, Little Rock, Arkansas
  - Synergy Research Center, Lemon Grove, California
  - Cenexel CNS, Los Alamitos, California
  - Cenexel RCA, Hollywood, Florida
  - Segal Trials, Miami Lakes, Florida
  - Cenexel ACMR, Atlanta, Georgia
  - Cenexel iResearch Atlanta, Decatur, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - Cenexel CBH, Gaithersburg, Maryland
  - Arch Clinical Trials, St Louis, Missouri
  - Cenexel HRI, Marlton, New Jersey
  - Neuro-Behavioral Clinical Research, North Canton, Ohio
  - Community Clinical Research, Austin, Texas

IPD SHARING:
Plan to Share IPD: No